CLINICAL TRIAL: NCT06840093
Title: Outcomes of Limited Postoperative Restrictions Following Sling Placement: A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Leanne E. Brechtel, Principle Investigator, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 202407515
Record Dates: First submitted 2025-02-06; First posted 2025-02-21 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Restriction; Midurethral Sling; Mesh; Stress Urinary Incontinence
Keywords: postoperative restrictions; midurethral sling; mesh; stress urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Limited Restrictions (Experimental): Patients will receive a handout with the following instructions:
  After discharge from the hospital, resume your normal activities as soon as you feel comfortable. There is no weight limit on lifting. There are no specific activities you should avoid (other than pelvic rest as described below).
  We recommend pelvic rest, nothing in the vagina (no intercourse, hot tubs, tub bathing or swimming) for 2 weeks. If you are prescribed vaginal estrogen, you may restart usage 1 week after surgery.
  A physical exam will be performed at your two-week appointment to check how your incision is healing. If there are no complications noticed at this appointment, there are no further pelvic restrictions. You can resume all activities, including vaginal intercourse, as tolerated.
  Interventions: Behavioral: Limited Restrictions
- Standard Restrictions (Active Comparator): Patient will receive a handout with the following instructions:
  After discharge from the hospital, avoid doing any strenuous activity (any activity that requires so much exertion that you cannot have a conversation comfortably while doing it).
  Do not lift anything over 15 pounds for 6 weeks after surgery. For 6 weeks, we recommend complete pelvic rest, nothing in the vagina (no intercourse, hot tubs, tub bathing or swimming). If you are prescribed vaginal estrogen, you may restart usage 1 week after surgery.
  A physical exam will be performed at your two-week appointment to check how your incision is healing.
  Interventions: Behavioral: Standard Restrictions

INTERVENTIONS:
Behavioral: Limited Restrictions — Patients will receive a handout with the following instructions: After discharge from the hospital, resume your normal activities as soon as you feel comfortable. There is no weight limit on lifting. There are no specific activities you should avoid (other than pelvic rest as described below). We recommend pelvic rest, nothing in the vagina (no intercourse, hot tubs, tub bathing or swimming) for 2 weeks.
  Arms: Limited Restrictions
Behavioral: Standard Restrictions — Patient will receive a handout with the following instructions: After discharge from the hospital, avoid doing any strenuous activity (any activity that requires so much exertion that you cannot have a conversation comfortably while doing it). Do not lift anything over 15 pounds for 6 weeks after surgery. For 6 weeks, we recommend complete pelvic rest, nothing in the vagina (no intercourse, hot tubs, tub bathing or swimming).
  Arms: Standard Restrictions

SUMMARY:
The purpose of this research study is to better understand optimal restrictions for patients postoperatively following a mesh urethral sling placement for patients with stress urinary incontinence.

Patients undergoing a midurethral sling procedure will be assigned to one of two groups. One group with be given standard postprocedural restrictions including instructions to avoid moderate activity and no lifting over 15lbs for six weeks after surgery. The other group will have fewer restrictions, with no restrictions on activity or lifting.

Participants will complete surveys at 2 weeks, 3 months and 1 year following their procedure to help providers better understand how patients are following postoperative restrictions and if there were any differences in the outcome of the procedure between the two groups.

DETAILED DESCRIPTION:
There is a growing body of evidence suggesting that strict postoperative restrictions may not be beneficial. Emerging data indicate that these restrictions do not significantly influence short- or long-term outcomes and may even have detrimental effects, such as increasing the incidence of venous thromboembolism and overall deconditioning.

Due to limited data on optimal postoperative restrictions following midurethral sling surgery, providers struggle to offer consistent, evidence-based recommendations. This variability can lead to inconsistent patient counseling, underscoring the need for further research to support or challenge universal postoperative restrictions.

Recent studies indicate that limited postoperative restrictions following pelvic organ prolapse surgery do not result in inferior outcomes. O'Shea et al. found that expedited activity post-surgery did not negatively affect anatomic or symptomatic results. Similarly, Mueller et al. reported that patients who resumed preoperative activities experienced fewer prolapse and urinary symptoms, with no inferior short-term anatomical outcomes. Arunachalam et al. also demonstrated that specific postoperative instructions did not significantly influence physical activity levels.

The latest guidelines for mesh hernia repair, the most common general surgery procedure involving synthetic mesh, recommend that patients resume activities without restriction post-surgery. Previous concerns that increased intra-abdominal pressure might lead to sling migration or mesh incorporation have not been substantiated. Studies show that abdominal pressures during daily activities overlap with those during physical exertion, and since patients cannot avoid daily activities like coughing or transitioning from sitting to standing, there is no physiological basis for strict restrictions.

While recent literature supports the safety of limited postoperative restrictions after pelvic prolapse surgery, this has not been validated for mid-urethral sling procedures. Traditionally, patients are advised to reduce activity for six to eight weeks post-surgery, which may deter physically active individuals from opting for the procedure. Given that the mid-urethral sling is considered the gold standard for treating stress urinary incontinence, relaxing restrictions and allowing quicker return to baseline activity could encourage more individuals to undergo this surgery.

Secondary Aims

* Compare incidence of adverse events, including mesh exposure, in each group
* Compare self-reported activity levels between groups
* Compare post-operative pain scores at 2 weeks and 3 months postoperatively
* Compare incidence of new onset dyspareunia

ELIGIBILITY:
Inclusion: Undergoing isolated synthetic mesh retropubic midurethral sling placement Exclusion criteria: Non-English speaking, incarcerated, cognitive impairment precluding informed consent, unable to ambulate without the assistance of an ambulation device, concurrent prolapse procedure

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Urogenital Distress Inventory | 3 months and 1 year postoperatively
  Questionnaire to assess the severity of lower urinary trat symptoms. Baseline compared to 3 months postoperatively with the hypothesis limited postoperative restrictions will result in non-inferior urinary symptoms compared to standard restrictions

SECONDARY OUTCOMES:
Incidence of adverse events | Primarily 3 months, will offer 1 year survey follow up
  All adverse events will be recorded for both groups
Self-reported activity | 2 weeks and 3 months postoperatively
  Using the Rapid Assessment of Physical Activity questionnaire, we will compare groups to assess if activity levels were different between the groups
Post-operative pain scores | 2 weeks and 3 months postoperatively
  Comparing post-operative pain scores at 2-weeks and 3-months post-operatively using the Numerical Pain Rating Scale from 0-10
Changes to Sexual Function | 3 months and 1 year postoperatively
  The Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-IR) will be administered at baseline, 3 months postoperatively and 1 year postoperatively to compare
Patient Impression of Improvement | 2 weeks, 3 months and 1 year postoperatively
  Using the Patient Global Impression of Improvement survey, will assess patient satisfaction and overall improvement

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Health Care, Iowa City, Iowa, United States